CLINICAL TRIAL: NCT06786130
Title: Burden and (Dis)Utility of Caregivers of Children With T1D
Brief Title: Societal Burden Associated With Type 1 Diabetes in Canada
Acronym: T1D
Status: Recruiting | Type: Observational
Sponsor: PeriPharm (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: BOD0250
Record Dates: First submitted 2024-09-16; First posted 2025-01-22 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes Mellitus; Quality of Life (QOL); Work Productivity; Caregiver Subjective Burden
Keywords: observational; quality of life; caregiver; work productivity; real-world
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Caregiver of child with T1D: Caregiver of child with T1D diagnosed within the past 2 years
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — This is an observational study in which participants complete PRO questionnaires via a web platform. No medical intervention or medication is involved.

SUMMARY:
The purpose of this observational study is to estimate the burden of T1D on caregivers of patient with T1D in terms of work productivity, healthcare resource utilization and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Parental caregiver of a child recently diagnosed (<= 2 years) with T1D before study inclusion;
2. Age ≥18 ;
3. Residence in the Canada;
4. Willingess to complete a 20-minute survey
5. Ability to read and understand French or English;
6. Signature of informed consent form (ICF)

Exclusion Criteria:

1. Participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parental caregivers of a child with T1D
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To estimate work productivity impairment of caregivers of a T1D child. | At recruitment
  Using the WOrk Productivity and Activity Impairment (WPAI) questionnaire

SECONDARY OUTCOMES:
To estimate healthcare resource utilization in caregivers of T1D child | At recruitment
  Using the modified Resource Utilization Questionnaire for Type 1 Diabetes (mRUQ-T1DM) questionnaire.
To estimate health-related quality of life in caregivers of a T1D child | At recruitment
  Using the EuroQOL-5 dimension-5 levels (EQ-5D-5L) questionnaire.
To estimate the caregiver burden in caregivers of a T1D child | At recruitment
  Using the Zarit Burden Interview-22 (ZBI-22) questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- PROxy Network, an initiative of PeriPharm Inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No